CLINICAL TRIAL: NCT06243510
Title: Comparison of Apixaban Versus Enoxaparin as Venous Thromboembolism Prophylaxis After Radical Cystectomy
Brief Title: Comparison of Apixaban Versus Enoxaparin
Acronym: CARE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: American Urological Association (Other)
Responsible Party: Principal Investigator, Katharine Michel, Resident, Abramson Cancer Center at Penn Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UPCC 15823
Record Dates: First submitted 2024-01-23; First posted 2024-02-06 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — apixaban; Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Enoxaparin (Active Comparator): Participants randomized to receive script for prophylactic dose of enoxaparin. Dosing will be done based on clinical providers (pharmacists) according to usual care. Participants will fill the script themselves.
  Interventions: Other: enoxaparin
- Apixaban (Experimental): Participants randomized to receive script for prophylactic dose of apixaban. Dosing will be done based on clinical providers (pharmacists) according to usual care. Participants will fill the script themselves.
  Interventions: Other: apixaban

INTERVENTIONS:
Other: apixaban — Participants will be randomized to receive a prescription for prophylactic apixaban
  Arms: Apixaban
Other: enoxaparin — Participants will be randomized to receive a prescription for prophylactic enoxaparin
  Arms: Enoxaparin

SUMMARY:
The goal of this randomized trial is to compare bladder cancer patient experiences taking prophylactic anticoagulation at home after surgery to remove their bladder. The main questions it aims to answer are:

* Are patients equally adherent to apixaban as they are enoxaparin? Why or why not?
* Do patients prefer apixaban or enoxaparin?
* What is the typical patient cost to take apixaban vs enoxaparin after surgery?

Participants will be randomized to receive a prescription for either enoxaparin or apixaban which they will then fill themselves and self-administer at home until post-operative day 30. They will receive phone calls from study coordinators at days 30 and 90 to complete questionaries over the phone to assess trial outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Able to communicate in English over the phone
4. Male or female, age >18 years
5. Diagnosed with biopsy-proven, urothelial cell carcinoma (any T stage, N0-1, M0) with plan for radical cystectomy with urinary diversion and concurrent pelvic lymph node dissection as treatment

Exclusion Criteria:

1. Preoperative use of a therapeutic dose of anticoagulant (this notably does not exclude patients taking antiplatelet agents)
2. Failure to undergo radical cystectomy with concurrent urinary diversion and pelvic lymph node dissection
3. Failure to be discharged by post-operative day 14
4. Failure to receive a script for enoxaparin or apixaban.
5. Any medical condition which precludes treatment with either enoxaparin or apixaban (including dialysis, hemophilia or any other bleeding diathesis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-11-24 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Adherence | Day of discharge to post-operative day 30
  proportion of days covered

SECONDARY OUTCOMES:
Cost | Day of discharge to post operative day 90
  patient out of pocket cost to fill their VTE prophylaxis prescription
Satisfaction as measured by 2. National Institute of Health (NIH) Patient-Reported Outcomes Measurement Information System (PROMIS) Medication Adherence Scale (PMAS) | Day of discharge to post-operative day 30
  patient satisfaction with their VTE prophylaxis drug
Reasons for non-adherence | Day of discharge to post-operative day 30
  patient-reported issues with adherence
VTE rate | Day of discharge to post-operative day 90
  rate of venous thromboembolism events
Bleeding rate | Day of discharge to post-operative day 90
  rate of major and minor bleeding events

CONTACTS AND LOCATIONS:
Overall Officials: Katharine F Michel, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-16): https://cdn.clinicaltrials.gov/large-docs/10/NCT06243510/Prot_SAP_000.pdf
  • Informed Consent Form (2024-01-16): https://cdn.clinicaltrials.gov/large-docs/10/NCT06243510/ICF_001.pdf